CLINICAL TRIAL: NCT06586333
Title: Evaluation of the Effect of an Education Program on Reducing the Efficacy and Costs of Inappropriate Stress Ulcer Prophylaxis in Intensive Care Units
Brief Title: Optimizing Stress Ulcer Prophylaxis Practices and Reducing Associated Costs in Intensive Care Units: a Nonrandomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Nilay Aksoy, Assoc.Professor, Altinbas University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/181
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stress Ulcer
Keywords: guidelines; adherence; stress ulcer; intensive care
MeSH Terms: conditions — Duodenal Ulcer | interventions — Pharmacists

STUDY DESIGN:
Intervention Model Description: Study Design and Participants The study is a prospectively designed, nonrandomized controlled study. It was conducted for six months at the EICU and GICU of a training and research hospital between 1 Jun 2023 and 1 December 2023.
  The study involved GICU patients as the standard care services observation group (OG). The use of SUP in the GICU was only monitored and noted. In the EICU, patients were identified as part of the recruiting guideline group (GG), and in addition to receiving usual care, they were managed for SUP according to the ASHP SUP guidelines [1]. The study duration was six months concurrently in the EICU and the GICU. Before inclusion, written informed consent was obtained from each patient or their parent(s)/legal guardian(s). Subjects with incomplete data were excluded. The inclusion criteria were patients aged ≥18 years and hospitalized for ≥24 hours in the EICU/GICU. Patients with a history of stomach cancer, admission to the ICU because of GI bleeding, subtotal/tot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Involved GICU patients as the standard care services observation group (OG). Stress ulcer prophylaxis were only observed and no intervention done
- Intervention (Experimental): In the EICU, patients were identified as part of the recruiting guideline group (GG), and in addition to receiving usual care, they were managed for SUP according to the ASHP stress ulcer prophylaxis guidelines
  Interventions: Drug: stress ulcer prophylaxis

INTERVENTIONS:
Drug: stress ulcer prophylaxis — In the EICU, patients were identified as part of the recruiting guideline group (GG), and in addition to receiving usual care, they were managed for SUP according to the ASHP SUP guidelines
  Other Names: clinical pharmacist
  Arms: Intervention

SUMMARY:
The study is a prospectively designed, nonrandomized controlled study. It was conducted for six months at the EICU and GICU of a training and research hospital between 1 Jun 2023 and 1 December 2023.

DETAILED DESCRIPTION:
The study involved GICU patients as the standard care services observation group (OG). The use of SUP in the GICU was only monitored and noted. In the EICU, patients were identified as part of the recruiting guideline group (GG), and in addition to receiving usual care, they were managed for SUP according to the ASHP SUP guidelines [1]. The study duration was six months concurrently in the EICU and the GICU. Before inclusion, written informed consent was obtained from each patient or their parent(s)/legal guardian(s). Subjects with incomplete data were excluded. The inclusion criteria were patients aged ≥18 years and hospitalized for ≥24 hours in the EICU/GICU. Patients with a history of stomach cancer, admission to the ICU because of GI bleeding, subtotal/total gastrectomy, or receiving a proton pump inhibitor for therapeutic purposes were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients aged ≥18 years and hospitalized for ≥24 hours in the EICU/GICU.

Exclusion Criteria:

* Patients with a history of stomach cancer, admission to the ICU because of GI bleeding, subtotal/total gastrectomy, or receiving a proton pump inhibitor for therapeutic purposes were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Adherence rates to ASHP guidelines | 6 months
  % of physician who adhere to ASHP guidelines

SECONDARY OUTCOMES:
Cost saving | 6 months
  The cost saving by adhere to ASHP guidelines

CONTACTS AND LOCATIONS:
Overall Officials: yunus emre Ayhan, Specialist clinical pharmacy, Study Chair — Prof. Dr. Cemil Taşcıoğlu City Hospital, Clinical Pharmacy, İstanbul, Türkiye,
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Clinical Pharmacy, İstanbul, Türkiye,, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No